CLINICAL TRIAL: NCT05104398
Title: Hemoperfusion With the Efferon CT Extracorporeal Adsorbers Containing Mesoporous Styrene-divinylbenzene Copolymer in Patients With Severe Covid-19
Brief Title: Hemoperfusion With the Efferon CT Extracorporeal Adsorbers in Patients With Severe Covid-19
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-ct-2021-02
Record Dates: First submitted 2021-10-31; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; mesoporous styrene-divinylbenzene copolymer; cytokines adsorption; hemoperfusion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline therapy: Group 1 (n=29) continued to receive standard treatment.
- Basic therapy + Efferon CT: group 2 (n=13) received HP procedure once, for 3-4 hrs, using Efferon CT adsorbers containing mesoporous SDC beads uptaking 6-60 kD molecules followed by continuous veno-venous hemodiafiltration. Group 2 included more severe patients requiring HP support.
  Interventions: Device: Efferon CT

INTERVENTIONS:
Device: Efferon CT — extracorporeal adsorbers containing mesoporous styrene-divinylbenzene copolymer to remove pro-inflammatory 6-60 kD molecules
  Groups: Basic therapy + Efferon CT

SUMMARY:
Direct extracorporeal removal of inflammatory mediators with various adsorbents has been suggested as a novel treatment modality for COVID-19 patients. Study determined safety, feasibility and effectiveness of clinical use of a hemoperfusion (HP) with a novel styrene- divinylbenzene copolymer (SDC) adsorbers to remove pro-inflammatory molecules from the bloodstream of COVID-19 patients.

DETAILED DESCRIPTION:
When a coronavirus is affected, the inflammatory process develops in a wide variety of organs and, in combination with a lack of oxygen, can lead to multiple organ failure. Acute respiratory distress syndrome (ARDS), seen in severe COVID-19, is characterized by shortness of breath and low blood oxygen levels. As a result, some patients may develop secondary bacterial and fungal infections. ARDS can lead to respiratory failure, which is the cause of death in 70% of COVID-19 deaths. In addition, the powerful release of cytokines by the immune system in response to viral infection and / or secondary infections can lead to symptoms of sepsis, which is the cause of death in 28% of COVID-19 cases, due to uncontrolled inflammation leading to multiple organ failure.

Most SARS-CoV patients who develop kidney failure end up dying. There is still no definitive answer to the question of why some COVID-19 patients are so severe - this may be partly due to concomitant diseases, although according to preliminary data from different countries it can be concluded that blocking the hyperactivation of immunity at the levels of IL-1 and IL- 6 may be effective in treating patients with severe coronavirus by suppressing or preventing cytokine storms.

Currently being treated COVID-19 is purely supportive. The main cause of death in seriously ill patients is acute respiratory failure. A possible reason for the development of this condition may be a cytokine storm, leading to acute decompensation of patients, which may be a possible direction of therapeutic intervention.

One of the main reasons for the high mortality rate of patients with the new coronavirus infection COVID-19 is the lack of etiotropic therapy. In this regard, pathogenetic therapy, aimed at key factors in the pathogenesis of emerging critical conditions, acquires great importance for saving the lives of patients.

Various pathogenetic treatment options are currently being discussed for the treatment of COVID-19, including selective inhibitors of various interleukins and extracorporeal cytokine elimination. So far, there is no convincing evidence of the effectiveness of the use of COVID-19 for any of them.

Nevertheless, according to many researchers, taking into account the peculiarities of pathogenesis, an important place in the pathogenetic treatment of patients with severe course of coronavirus infection should be occupied by methods of extracorporeal hemocorrection. They have complex multiple effects and can quickly normalize the level of cytokines and other factors of pathogenesis and thereby prevent or reduce the severity of organ disorders.

When planning this clinical trial, it was suggested that hemosorption of cytokines could improve outcome in critically ill COVID-19 patients with suspected cytokine storms.

Hemosorption device Efferon CT provides a decrease in high concentrations of endogenous mediators of the systemic inflammatory response, incl. cytokines leading to the development of multiple organ failure and other pathophysiological disorders. The device for hemosorption Efferon CT has a high adsorption capacity and biocompatibility.

Efferon CT (Efferon JSC, Moscow, Russia) - a device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by removing excess cytokines, myoglobin, endogenous and exogenous toxic substances from the patient's blood.

Efferon СT is a cylindrical polycarbonate body filled with spherical granules of a polymeric cross-linked porous hemosorbent based on a hypercrosslinked styrene-divinylbenzene copolymer and isotonic sodium chloride solution.

The device is manufactured according to TU 32.50.50-001-12264678-2018, passed the necessary tests and is registered in Russia as a medical device RZN 2019/8886.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 21-80,
* Primary ICU patients (admitted to the hospital, transfer from another hospital or department less than 72 hours),
* Positive PCR test for SARS-CoV-2,
* PaO2 / FiO2 <300,
* SOFA ≥ 4 with clinic of organ dysfunction.

Exclusion Criteria:

* Pregnancy,
* The presence of signs of a bacterial infection or the addition of secondary purulent-septic complications,
* Cancer (including blood diseases),
* Chronic diseases in the stage of decompensation,
* Recent or ongoing bleeding,
* Syndrome of disseminated intravascular coagulation,
* Thrombocytopenia,
* Patients in terminal condition or receiving palliative care,
* Patients for whom, for any reason, the use of anticoagulants is not safe.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 42 COVID-19, PCR+ patients, age <81 years, average 63 (SD range, 54-69) years, 52% men
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon CT hemoperfusion on pulmonary oxygen metabolism function | 1-120 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 120 hours

SECONDARY OUTCOMES:
Effect of Efferon CT hemoperfusion on SOFA scores | 1-120 hours
  Value of indicators on the SOFA scale every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 120 hours
Effect of Efferon CT hemoperfusion on IL-6 levels | 1-120 hours
  Value of IL-6 levels from the start of hemoperfusion (hour 0) to 120 hours
Effect of Efferon CT hemoperfusion on Ferritin levels | 1-120 hours
  Value of Ferritin levels from the start of hemoperfusion (hour 0) to 120 hours
Effect of Efferon CT hemoperfusion on Lactate levels | 1-120 hours
  Value of Lactate levels from the start of hemoperfusion (hour 0) to 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Timur Kim, MD, Principal Investigator — N.I. Pirogov Clinical City Hospital No. 1
Locations (1):
- N.I. Pirogov City Clinical Hospital No. 1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco C, Bagshaw SM, Bellomo R, Clark WR, Husain-Syed F, Kellum JA, Ricci Z, Rimmele T, Reis T, Ostermann M. Extracorporeal Blood Purification and Organ Support in the Critically Ill Patient during COVID-19 Pandemic: Expert Review and Recommendation. Blood Purif. 2021;50(1):17-27. doi: 10.1159/000508125. Epub 2020 May 26. PMID 32454500
- [Background] Ronco C, Reis T, De Rosa S. Coronavirus Epidemic and Extracorporeal Therapies in Intensive Care: si vis pacem para bellum. Blood Purif. 2020;49(3):255-258. doi: 10.1159/000507039. Epub 2020 Mar 13. No abstract available. PMID 32172242
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578